CLINICAL TRIAL: NCT03236766
Title: Engaging Pacific Islander Perspectives on Mental Illness and Mental Health Services
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No intervention or clinical trial necessitating participants ultimately needed or required for this study.
Sponsor: University of California, Riverside (Other)
Responsible Party: Principal Investigator, Andrew Subica, Assistant Professor, University of California, Riverside
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R21MH110814 (NIH)
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No intervention (Other)
  Interventions: Other: Citizens' panels

INTERVENTIONS:
Other: Citizens' panels — This study is exploratory in nature, designed to capture lay Pacific Islanders' thoughts and beliefs about existing service engagement approaches. Therefore, there are no study arms to list.

SUMMARY:
This study will enroll 100 Samoan and 100 Marshallese adults to discuss mental health, mental disorders, and approaches for engaging Pacific Islander adults with mental illness into mental health services.

DETAILED DESCRIPTION:
Despite enduring high mental health burden, Pacific Islanders have received minimal research or clinical attention in the US. Due to our poor understanding of the issues surrounding Pacific Islander mental health, engaging Pacific Islanders in mental health services has been very difficult.

This study draws from the Cultural Determinants of Help-Seeking Model to address this research and clinical gap by conducting focus groups and citizens' panels to obtain public input from 50 Samoans in LAC and 50 Marshallese in Arkansas on their unique mental health perspectives, needs, barriers and facilitators to services, and strategies to overcome these barriers. The citizens' panels will bring together lay public members, present multiple viewpoints about various mental health issues, and have members deliberate and reach a collective decision on these issues. All group materials will be translated into English, Samoan, and Marshallese, and interpreters will be present during the sessions. The groups will be audio-recorded, transcribed verbatim, and analyzed by the Research Team for themes. Numerical data will also be collected about levels of public awareness about mental illness, mental health stigma, acculturation, and underutilization of mental health services from 100 Samoan and 100 Marshallese community members to better understand these possible service barriers.

Analyzed data will be used to develop a set of intervention components that are likely to increase service engagement among both Samoans and Marshallese. These components will provide the foundation for a universal service engagement intervention for Pacific Islanders that will be developed and tested in future research.

ELIGIBILITY:
Inclusion Criteria:

* Samoan or Marshallese heritage; living in Los Angeles County or Northwest Arkansas; age 18 years or older; English, Samoan, or Marshallese oral and reading fluency

Exclusion Criteria:

* Not of Samoan or Marshallese heritage; living outside the catchment areas; younger than 18 years; not fluent in English, Samoan, or Marshallese

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants participating in study | Up to 20 months
  There is no primary quantitative outcome beyond increased knowledge of Pacific Islander mental health beliefs and treatment preferences

IPD SHARING:
Plan to Share IPD: No